CLINICAL TRIAL: NCT04796064
Title: Comparative Effectiveness Study of Low Versus High-Intensity Aerobic Training in Community-dwelling Older Men With Post-COVID 19 Sarcopenia
Brief Title: Low Versus High-Intensity Aerobic Training in Community-dwelling Older Men With Post-COVID 19 (SARS-CoV-2) Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Eid, assistant professor of physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sarcopenia
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-intensity aerobic training group (Experimental)
  Interventions: Other: low-intensity aerobic training
- high-intensity aerobic training group (Experimental)
  Interventions: Other: low-intensity aerobic training

INTERVENTIONS:
Other: low-intensity aerobic training — A low-intensity aerobic training group started with 15 minutes of warm-up, which includes static stretching of the upper and lower limb muscles. then participants were instructed to do 30 minutes of low-intensity aerobic training exercises, which include 20 minutes on the treadmill and 10 minutes of cycle ergometer, followed by 10 minutes of cool down.
  - In high-intensity training (HAT) the same protocol has been followed, but the intensity of exercises was fixed between 60% to 80 % of maximum heart rate. The strength training includes major group muscles such as shoulder flexors, extensors, and abductors, elbow flexors and extensors, hip flexors& extensors, knee flexors&extensors, abdominal and back muscles also were trained. Each group of muscles was trained for 10 repetitions for 3 sets with a rest period of 5 minutes.

SUMMARY:
Sarcopenia is the major health concern and common consequence of COVID-19 in the ageing population. The objective of this study is to find and compare low and high-intensity aerobic training protocols on clinical and psychological effects in community-dwelling older men with post-COVID 19 Sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 60 - 80 years with
* A positive diagnosis of post-COVID-19 sarcopenia

Exclusion Criteria:

* Under medication
* History of lower limb surgeries, fractures
* Cardiac problems
* Respiratory problems
* Neurological problems
* Systemic problems and any other contraindications for aerobic training

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Handgrip strength | 8 weeks
  It is a simple and cost-effective test to measure the upper limb strength

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Eid, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided